CLINICAL TRIAL: NCT02191891
Title: A Phase Ib Open-label Clinical Trial of Once Daily Oral Treatment of Afatinib Plus Weekly Intravenous Infusion of Xentuzumab (BI 836845) in Patients With EGFR Mutant Non-small Cell Lung Cancer With Progression Following Prior EGFR Tyrosine Kinase Inhibitors
Brief Title: Xentuzumab (BI 836845) Plus Afatinib in Patients With Epidermal Growth Factor Receptor (EGFR) Mutant Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1280.16
Record Dates: First submitted 2014-07-14; First posted 2014-07-16 (Estimated); Results first posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — xentuzumab; Afatinib

ARMS (5):
- Xentuzumab + Afatinib 30 milligram (mg) - Part A (Experimental): Patients received intravenous infusion of Xentuzumab 1000 milligram (mg) delivered over 60 minutes per week for 4 weeks, in combination with once daily oral treatment of Afatinib 30 mg film-coated tablet. Dose confirmation part (Part A).
  Interventions: Drug: Xentuzumab; Drug: Afatinib
- Xentuzumab + Afatinib 40 mg - Part A (Experimental): Patients received intravenous infusion of Xentuzumab 1000 milligram (mg) delivered over 60 minutes per week for 4 weeks, in combination with once daily oral treatment of Afatinib 40 mg film-coated tablet. Dose confirmation part (Part A).
  Interventions: Drug: Xentuzumab; Drug: Afatinib
- Xentuzumab + Afatinib 20 mg - Part B (Experimental): Patients received intravenous infusion of Xentuzumab 1000 milligram (mg) delivered over 60 minutes per week for 4 weeks, in combination with once daily oral treatment of Afatinib 20 mg film-coated tablet. Expansion part (Part B).
  Interventions: Drug: Xentuzumab; Drug: Afatinib
- Xentuzumab + Afatinib 30 mg - Part B (Experimental): Patients received intravenous infusion of Xentuzumab 1000 milligram (mg) delivered over 60 minutes per week for 4 weeks, in combination with once daily oral treatment of Afatinib 30 mg film-coated tablet. Expansion part (Part B).
  Interventions: Drug: Xentuzumab; Drug: Afatinib
- Xentuzumab + Afatinib 40 mg - Part B (Experimental): Patients received intravenous infusion of Xentuzumab 1000 milligram (mg) delivered over 60 minutes per week for 4 weeks, in combination with once daily oral treatment of Afatinib 40 mg film-coated tablet. Expansion part (Part B).
  Interventions: Drug: Xentuzumab; Drug: Afatinib

INTERVENTIONS:
Drug: Xentuzumab — Patients received intravenous infusion of Xentuzumab 1000 milligram (mg) delivered over 60 minutes per week for 4 weeks, in combination with once daily oral treatment of Afatinib film-coated tablet.
  Other Names: BI 836845
Drug: Afatinib — Patients received intravenous infusion of Xentuzumab 1000 milligram (mg) delivered over 60 minutes per week for 4 weeks, in combination with once daily oral treatment of Afatinib film-coated tablet.

SUMMARY:
Part A: To determine the maximum tolerated dose (MTD) and/or recommended phase II dose (RP2D) of Xentuzumab (BI 836845) in combination with afatinib in patients with non-small cell lung cancer with progression following prior treatment (EGFR TKI or platinum-based chemotherapy).

Part B: To evaluate the early anti-tumour activity of Xentuzumab (BI 836845) in combination with afatinib in patients with EGFR mutant non-small cell lung cancer with progression following prior irreversible EGFR TKIs.

Part A and B: To evaluate the safety and pharmacokinetics of BI 836845 in combination with afatinib in patients with non-small cell lung cancer

ELIGIBILITY:
Inclusion criteria:

* Aged 18 years or older
* Pathologically confirmed of advanced and/or metastatic stage IIIb/IV non-small cell carcinoma of lung
* Activating EGFR mutation (exon 19 deletion, L858R, G719X, L861X)
* Presence of EGFR activating mutation and absence of EGFR T790M in the tumour associated with the latest disease progression. Only applicable in Part B
* Must have adequate fresh or archival tumour tissue at the late disease progression immediately prior to the study entry
* Part A: Progression of disease (RECIST 1.1) while on continuous treatment with single EGFR TKI or for histology other than adenocarcinoma and without prior EGFR TKI treatment: progression of disease (RECIST v1.1) on platinum-based chemotherapy. Part B: Progression of disease (RECIST v1.1) while on continuous treatment with single agent of the second generation irreversible EGFR TKI (e.g. afatinib or dacomitinib)
* No intervening systemic therapy between cessation of EGFR TKI and study treatment
* Patient must have measurable disease per RECIST 1.1 presented after tumour biopsy for the late disease progression
* Eastern Cooperative Oncology Group (ECOG) performance score 0 or 1
* Life expectancy of >= 3 months
* Fasting plasma glucose < 8.9 mmol/L (< 160mg/dL) and HbA1C < 8%
* Adequate organ function
* Recovered from any previous therapy related toxicity to <= Grade 1 at study entry (except for stable sensory neuropathy <= Grade 2 and alopecia)
* Written informed consent that is consistent with ICH-GCP guidelines and local regulations
* No known potentially targetable mutation other than IGF signaling pathway or EGFR or no available treatment for potentially targetable mutation

Exclusion criteria:

* Part A only: For patient who has been treated with afatinib: last treatment at reduced dose below the assigned dose level
* Patient whose disease progressed on insufficient dose of EGFR TKI immediately prior to study in the opinion of the investigator
* More than 2 prior EGFR TKI treatment regimens for Part B
* Chemotherapy, biological therapy or investigational agents (except EGFR TKIs) within 4 weeks
* Use of previous EGFR TKIs except afatinib within 3 days
* Radiotherapy within 4 weeks prior to the start of study treatment
* Active brain or subdural metastases
* Meningeal carcinomatosis.
* Major surgery (as judged by the investigator) within 4 weeks
* Known hypersensitivity to afatinib, monoclonal antibody
* Prior severe infusion-related reaction to a monoclonal antibody
* History or presence of clinically relevant cardiovascular abnormalities
* Female patients of childbearing potential (see Section 4.2.2.3) and male who are able to father a child
* Any history of or concomitant condition that, in the opinion of the investigator not to comply with the study or interfere with the evaluation of the efficacy and safety of the test drug
* Previous or concomitant malignancies at other sites, except effectively treated non-melanoma skin cancers, carcinoma in situ of the cervix, ductal carcinoma in situ or effectively treated malignancy that has been in remission for more than 3 years and is considered to be cured.
* Disease that is considered by the investigator to be rapidly progressing or life threatening such as extensive symptomatic visceral disease including hepatic involvement and pulmonary lymphangitic spread of tumour (subjects who are intended for urgent chemotherapy)
* Requiring treatment with any of the prohibited concomitant medications
* Known pre-existing interstitial lung disease (ILD)
* Any history or presence of poorly controlled gastrointestinal disorders that could affect the absorption of the study drug
* Active hepatitis B infection active hepatitis C infection and/or known HIV carrier.
* Previous treatment with agents targeting the insulin like growth factor (IGF) signalling pathway.
* Previous treatment with EGFR TKI which cannot be documented as either reversible or irreversible (Part B only)
* Part B only: Prior treatment with third generation irreversible EGFR TKI (e.g. AZD9291 or CO-1686)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-10-21 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (10):
- National Hospital Organization Kyushu Cancer Center, Fukuoka, Fukuoka, Japan
- National Cancer Centre Singapore, Singapore, Singapore
- South Korea (4):
  - Chungbuk National University Hospital, Cheongju-si
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
- Taiwan (4):
  - Chang Gung Memorial Hospital Chiayi, Chiayi City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - NCKUH, Tainan
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'.
  For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with epidermal growth factor receptor (EGFR) mutant lung cancer were recruited in this multi-centre, open-label, phase Ib clinical trial. The trial consisted of a dose confirmation part (Part A) and an expansion cohort (Part B), where Part A and Part B were conducted sequentially.
Pre-assignment Details: All patients were screened for eligibility to participate in the trial. Patients attended specialist sites which would then ensure that they (all patients) met all inclusion/exclusion criteria. Patients were not to be entered to trial treatment if any one of the specific entry criteria were not met.
Period: Overall Study
Arm/Group | Xentuzumab + Afatinib 30 Milligram (mg) - Part A | Xentuzumab + Afatinib 40 mg - Part A | Xentuzumab + Afatinib 20 mg - Part B | Xentuzumab + Afatinib 30 mg - Part B | Xentuzumab + Afatinib 40 mg - Part B
Started | 4 | 12 | 4 | 2 | 10
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 12 | 4 | 2 | 10
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 2
Not completed — Disease Progression | 4 | 10 | 4 | 2 | 7

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This patient set included all patients who were documented to have received and taken at least 1 dose of any study drug during the treatment courses (from Day 1).
Groups:
- Total: Total of all reporting groups
Arm/Group | Xentuzumab + Afatinib 30 Milligram (mg) - Part A | Xentuzumab + Afatinib 40 mg - Part A | Xentuzumab + Afatinib 20 mg - Part B | Xentuzumab + Afatinib 30 mg - Part B | Xentuzumab + Afatinib 40 mg - Part B | Total
Number analyzed (Participants) | 4 | 12 | 4 | 2 | 10 | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.75 (9.11) | 59.08 (10.16) | 57.75 (9.5) | 68.00 (2.83) | 56.60 (9.94) | 59.03 (9.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 2 | 0 | 8 | 17
  Male | 2 | 7 | 2 | 2 | 2 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 12 | 4 | 2 | 10 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 12 | 4 | 2 | 10 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Dose Limiting Toxicities (DLT) - Part A
Description: DLT Criteria: Common Terminology Criteria for Adverse Events(CTCAE) CTCAE Grade (G) 4 neutropenia lasting ≥7 days; Febrile neutropenia with a single/sustained temperature of ≥38.3°C for >1 hour; Documented infection with absolute neutrophil count (ANC) <1.0 x 109/L; G 3/4 thrombocytopenia associated with bleeding requiring platelet transfusion; G 2/higher decrease in cardiac left ventricular function; G 2 diarrhea lasting for ≥7 days; G ≥3 diarrhea; G≥3 nausea/vomiting; G≥3 skin rash; aspartate aminotransferase (AST)/alanine aminotransferase (ALT) >5 x Upper limit of normal (ULN)/>baseline value +4 x ULN; G≥3 fatigue/asthenia lasting for >7 days; G≥3 hyperglycemia lasting >48 hours; All other non-hematologic adverse events(AEs) of G≥3 (except alopecia, infusion reaction, and allergic reaction) that led to an interruption of afatinib/xentuzumab for >14 days until recovery to baseline/G 1; Any other study drug-related toxicity considered significant enough to qualify as DLT.
Time Frame: During the first treatment course, up to 28 days.
Population: Maximum Tolerated Dose (MTD) Set (MS): this patient set defined the set of patients in Part A who were fully evaluable for determination of the MTD in the first treatment course.
Measure: Number; unit: Participants
Arm/Group | Xentuzumab + Afatinib 30 Milligram (mg) - Part A | Xentuzumab + Afatinib 40 mg - Part A
Number analyzed (Participants) | 3 | 12
Participants | 0 | 0

2. Primary Outcome: Maximum Tolerated Dose (MTD) - Part A
Description: Maximum tolerated dose (MTD) of Xentuzumab in combination with Afatinib, in patients with non-small cell lung cancer with progression following prior treatment, based on the occurrence of dose limiting toxicity (DLT) during the first treatment course. MTD was defined as the highest dose level examined of trial medication, at which no more than 1 out of 6 patients experienced a DLT during the MTD evaluation period.
Time Frame: During the first treatment course, up to 28 days.
Population: as for outcome 1
Measure: Number; unit: Milligrams (mg)
Groups:
- Xentuzumab + Afatinib - Part A: In the dose-escalation phase patients received intravenous infusion of Xentuzumab 1000 milligram (mg) delivered over 60 minutes per week for 4 weeks, in combination with once daily oral treatment of Afatinib 30/40 mg film-coated tablet until the patient met criteria for stopping study medication during the MTD evaluation period.
Arm/Group | Xentuzumab + Afatinib - Part A
Number analyzed (Participants) | 15
Milligrams (mg) | 40

3. Primary Outcome: Number of Participants With Objective Response (OR) - Part B
Description: OR was defined as best overall response of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumours (RECIST) v1.1, where best overall response was defined according to RECIST v1.1 from first administration of trial medication until the earliest of disease progression, death or last evaluable tumour assessment before start of subsequent anti-cancer therapy.
Time Frame: Tumour assessment was performed every 4 weeks after the start of treatment for first 8 weeks, in 8-week intervals thereafter and in 12-week interval after Course 16 until disease progression or the start of further anti-cancer treatment, up to 1200 days.
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | Xentuzumab + Afatinib 20 mg - Part B | Xentuzumab + Afatinib 30 mg - Part B | Xentuzumab + Afatinib 40 mg - Part B
Number analyzed (Participants) | 4 | 2 | 10
Participants | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Disease Control (DC) - Part B
Description: DC was defined as best overall response of complete response (CR) or partial response (PR) or stable disease (SD) according to RECIST v1.1, where best overall response was defined according to RECIST v1.1 from first administration of trial medication until the earliest of disease progression, death or last evaluable tumour assessment before start of subsequent anti-cancer therapy.
Time Frame: as for outcome 3
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | Xentuzumab + Afatinib 20 mg - Part B | Xentuzumab + Afatinib 30 mg - Part B | Xentuzumab + Afatinib 40 mg - Part B
Number analyzed (Participants) | 4 | 2 | 10
Participants | 2 | 2 | 6

5. Secondary Outcome: Time to OR - Part B
Description: Time to OR, defined as the time from first treatment administration until first documented CR or PR. For patients with OR, time to OR was summarised on a patient level.
Time Frame: as for outcome 3
Population: TS - Patients with objective response (There were no patients with objective response in the expansion cohort)
Arm/Group | Xentuzumab + Afatinib 20 mg - Part B | Xentuzumab + Afatinib 30 mg - Part B | Xentuzumab + Afatinib 40 mg - Part B
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Duration of OR - Part B
Description: Duration of OR, defined as the time from first documented CR or PR until the earliest of disease progression or death among patients with OR - Part B. For patients with OR, duration of OR was summarised on a patient level.
Time Frame: as for outcome 3
Population: TS - Patients with objective response (There were no patients with objective response in the expansion cohort)
Arm/Group | Xentuzumab + Afatinib 20 mg - Part B | Xentuzumab + Afatinib 30 mg - Part B | Xentuzumab + Afatinib 40 mg - Part B
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first administration of trial medication until end of the follow-up period, up to 1247 days.
Description: Treated set (TS): This patient set included all patients who were documented to have received and taken at least 1 dose of any study drug during the treatment courses (from Day 1).
  As per protocol safety data was collected according to dose groups.
Groups:
- Xentuzumab + Afatinib 20 mg: Patients received intravenous infusion of Xentuzumab 1000 mg delivered over 60 minutes per week for 4 weeks, in combination with once daily oral treatment of Afatinib 20 mg film-coated tablet.
- Xentuzumab + Afatinib 30 mg: Patients received intravenous infusion of Xentuzumab 1000 mg delivered over 60 minutes per week for 4 weeks, in combination with once daily oral treatment of Afatinib 30 mg film-coated tablet.
- Xentuzumab + Afatinib 40 mg: Patients received intravenous infusion of Xentuzumab 1000 mg delivered over 60 minutes per week for 4 weeks, in combination with once daily oral treatment of Afatinib 40 mg film-coated tablet.
Arm/Group | Xentuzumab + Afatinib 20 mg | Xentuzumab + Afatinib 30 mg | Xentuzumab + Afatinib 40 mg
All-Cause Mortality (participants affected / at risk) | 0/4 | 1/6 | 2/22
Serious Adverse Events (participants affected / at risk) | 0/4 | 2/6 | 8/22
Other Adverse Events (participants affected / at risk) | 4/4 | 6/6 | 20/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Xentuzumab + Afatinib 20 mg (N=4) | Xentuzumab + Afatinib 30 mg (N=6) | Xentuzumab + Afatinib 40 mg (N=22)
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Xentuzumab + Afatinib 20 mg (N=4) | Xentuzumab + Afatinib 30 mg (N=6) | Xentuzumab + Afatinib 40 mg (N=22)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 16
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 3
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 4 | 2
Tongue ulceration (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2
Chest pain (General disorders) | 0 | 0 | 2
Fatigue (General disorders) | 1 | 0 | 4
Mucosal inflammation (General disorders) | 0 | 0 | 5
Oedema peripheral (General disorders) | 0 | 0 | 3
Pain (General disorders) | 0 | 1 | 0
Xerosis (General disorders) | 0 | 1 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 2
Paronychia (Infections and infestations) | 1 | 2 | 11
Rash pustular (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 2
White blood cell count decreased (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 3
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Nail dystrophy (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3 | 5
Rash (Skin and subcutaneous tissue disorders) | 2 | 3 | 10
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-11-02): https://cdn.clinicaltrials.gov/large-docs/91/NCT02191891/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-27): https://cdn.clinicaltrials.gov/large-docs/91/NCT02191891/SAP_001.pdf